CLINICAL TRIAL: NCT00425243
Title: Evaluation of the Long-Term Efficacy and Safety of Zolpidem-MR 12.5 mg Compared to Placebo, When Both Are Administered Over a Long-Term Period "as Needed", in Patients With Chronic Primary Insomnia
Brief Title: Efficacy and Safety of Zolpidem-MR Administered Over a Long Term Period as Needed for Insomnia (ZOLONG)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Sanofi (Industry)
Responsible Party: ICD Study Director, sanofi-aventis
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: LTE5407
Record Dates: First submitted 2007-01-19; First posted 2007-01-22 (Estimated); Last update posted 2009-04-06 (Estimated); Status verified 2009-04

CONDITIONS: Sleep Initiation and Maintenance Disorders
Keywords: primary insomnia; chronic insomnia
MeSH Terms: conditions — Sleep Initiation and Maintenance Disorders

STUDY DESIGN:
Who Masked: Participant, Investigator

INTERVENTIONS:
Drug: zolpidem-MR (SL800750)

SUMMARY:
The primary objective of the study is to evaluate the hypnotic efficacy of zolpidem-MR 12.5 mg in comparison with placebo, when administered over a long-term period, on an "as needed" basis, in patients with chronic primary insomnia.

Secondary objectives of the study are to evaluate the drug taking behavior over a long-term period and the clinical safety and tolerability of zolpidem-MR 12.5 mg in comparison to placebo administered over a long-term period, on an as needed basis.

ELIGIBILITY:
Inclusion Criteria:

* patients with chronic primary insomnia

The investigator will evaluate whether there are other reasons why a patient may not participate.

Ages: 18 Years to 64 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 1025 (Actual)
Dates: Start 2004-08; Primary Completion 2006-01 (Actual); Study Completion 2006-01 (Actual)

PRIMARY OUTCOMES:
The primary efficacy variable is item 1 (which assessed sleep aid) of the Patient Global Impression (PGI) scale at week 12.

SECONDARY OUTCOMES:
Main secondary variables are the Clinical Global Impression (CGI) improvement item and to items 2, 3, and 4 of the PGI scale at week 12.

CONTACTS AND LOCATIONS:
Overall Officials: ICD CSD, Study Director — Sanofi
Locations (1):
- Sanofi-Aventis, Malvern, Pennsylvania, United States

REFERENCES:
- [Result] Krystal AD, Erman M, Zammit GK, Soubrane C, Roth T; ZOLONG Study Group. Long-term efficacy and safety of zolpidem extended-release 12.5 mg, administered 3 to 7 nights per week for 24 weeks, in patients with chronic primary insomnia: a 6-month, randomized, double-blind, placebo-controlled, parallel-group, multicenter study. Sleep. 2008 Jan;31(1):79-90. doi: 10.1093/sleep/31.1.79. PMID 18220081